CLINICAL TRIAL: NCT03974646
Title: Effectiveness of Chronic Kidney Disease Nurse-led Self-management Program (CKD-NLSM): A Randomized Controlled Trial.
Brief Title: Effectiveness of Chronic Kidney Disease Nurse-led Self-management Program (CKD-NLSM)
Acronym: CKD-NLSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Boon-How Chew, Associate Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAlSawad
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Renal Insufficiency
Keywords: chronic kidney disease; health related quality of life; knowledge; randomized controlled trial; self-management; self-efficacy; social cognitive theory
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: patients fulfilling eligibility criteria and willing to participate will randomized after baseline assessment (1:1 allocation ration). A prior, an independent research assistant will prepare a computer-generated randomization schedule. The allocation numbers will be concealed in opaque sealed envelopes prepared by a research assistant. the envelopes will be accessible by the research assistant, only opening them after informed consent and baseline assessment have been obtained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants assigned to the intervention group will receive both will receive usual care (standard clinical and medical services) provided to individual with CKD stages 3-4 who attend the CKD clinic at medical outpatient department on their clinic follow up , and a 12- weeks self-management intervention delivered by two dedicated and trained renal nurse educators. The intervention will involve three group-based sessions, CKD booklet and three follow-up phone calls.
  Interventions: Behavioral: Nurse-led self-management Program
- control group (No Intervention): Participants randomized to the control group in this study will receive usual care (standard clinical and medical services) provided to individual with CKD stages 3-4 who attend the CKD clinic at medical outpatient department on their clinic follow up. Usual care consisted of brief verbal information (2-5 minutes) about taking medications, reducing salt, smoking cessation and reducing alcohol consumption. There will no structured program but only the provision of written material to patients.

INTERVENTIONS:
Behavioral: Nurse-led self-management Program — Group-based sessions will be scheduled at week two, week four and week six. Participant will be given a printed booklet Participants will receive three individual follow-up phone calls of 20-30 minutes each at week three, week five and week seven.
  Arms: intervention group

SUMMARY:
This study aims to develop, implement and evaluate the effectiveness of a theory-driven nurse-led self-management intervention program compared to standard usual care in people with CKD stages 3-4 on CKD knowledge, self-management behavior, self-efficacy and HRQoL using valid and reliable instruments in Malaysia.

DETAILED DESCRIPTION:
Patients aged ≥ 18 years with CKD stages 3-4 will be recruited between July 2019 - October 2019. Participants will be randomly allocated into either the intervention (N = 77) or control group (N = 77). The control group will receive standard usual care, while the intervention group will receive standard usual care plus a self-management program delivered by renal nurse educators. The intervention will be guided by social cognitive theory and include group-based educational sessions, CKD booklet and follow-up phone calls. Both groups will be followed for 12 weeks. Data will be analyzed using SPSS version 25. The primary outcomes are improving in knowledge and self-management, while the secondary outcomes are improving in self-confidence, quality of life and clinical outcomes of the participants.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are CKD (stages 3-4), aged ≥ 18 years, could speak, read, and understand Malay language, able to give informed consent, had never participated in any structured education program before, willing to participate in the study and most importantly not expected to start dialysis during the study.

Exclusion Criteria:

* Participants will be excluded if they had ESRD, were receiving dialysis or were cognitively impaired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change CKD knowledge | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  kidney disease knowledge will be measured using a self-report instrument Kidney Disease Knowledge Survey (KiKS). It includes 28 questions, 5 multiple choice type questions and 23 Yes-No questions; none of the questions included an "I don´t know" option. To assess the survey score, 1 point was given to each correct answer and zero to each wrong one. The questionnaire doesn't have domains, and the total score was calculated as the sum of the correct responses to each question divided by the total number of questions, which results in values from 0 to 1 where 1 means the highest level of knowledge.
Change CKD Self-Management Behavior | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  CKD self-management behavior will be assessed by Self-report instrument Chronic Kidney Disease Self-management (CKD-SM) by (C. C. Lin et al., 2013). CKD-SM instrument contains of 29-item to measure participants' self-management behavior factors. Each item is scored on a Likert scale from 1-4 with 1 being 'never' and 4 'always'. Total scores of the CKD-SM range from 29 to 116 and higher scores indicate better self-management behavior in managing CKD.

SECONDARY OUTCOMES:
Change Self-efficacy to manage CKD. | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  Self-efficacy will be measured by using a self-report instrument the Stanford Self-Efficacy for Managing Chronic Disease - 6-item Scale. This widely used six-item instrument was derived from several self-efficacy scales developed and tested for the Chronic Disease Self-Management study by Lorig et al., 2001. Each item is scored on a 10-point Likert scale ranging from "not at all confident" (1) to "totally confident" (10), with a total score ranging from 6-60. The scale is scored by calculating the mean of at least four of the six items, therefore allowing for a maximum of two missing items. A higher number indicates a higher self-efficacy.
Change Health-related quality of life (HRQoL): Malay KDQOL-36TM | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  Health-related quality of life will be assessed using a self-report instrument Malay version of the Kidney Disease Quality of life (KDQOL-36TM) originally developed by RAND Health Organization, the University of Arizona for individuals with CKD and on dialysis. KDQOL-36TM consists of 12 items which measure physical functioning (physical component summary PCS) and mental functioning (mental component summary MCS), four items to assess the burden of kidney disease, 12 items for symptoms and problems, and eight items to measure the effects of kidney disease on daily life. The scores of the KDQOL-36TM are transformed into 0 to 100, with higher scores indicating better HRQoL.
Change Systolic Blood Pressure | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  Systolic Blood Pressure will be assessed using CARESCAPE DINAMAP technology digital blood pressure monitor model V100, BP assessor will obtain three BP measures in the right arm after the participant has been sitting quietly for 5 min. An average of the 3 measures is recorded. The recommended Systolic Blood Pressure lower of 130 mm Hg.
Change 24-hour Urine Creatinine | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  24-hour urine creatinine will assessed using Jaffe, rate blanking for 24 hour urine collection with (mmol/24Hr) units of measures. The reference range for Males:3.45-21 mmol/24h and for Females: 7-14 mmol/24h. Higher than 21 mmol/24h and higher thank 14 mmol/24h is not recommended for male and female respectively.
Change 24-hour Urine Protein | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  24-hour urine protein will assessed using Turbidimetric method Benzethonium chloride for 24 hour urine collection with (g/24Hr) units of measures. The reference range <0.14 g/24h. Higher than<0.14 g/24h is not recommended.
Change 24-hour Urine Urea | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  24-hour Urine Urea will assessed using Kinetic test with urease and glutamate dehydrogenase for 24 hour urine collection with (mmol/24Hr) units of measures. The reference range is 428-714 mmol/24h. Higher than 714 mmol/24h is not recommended.
Change 24-hour Urine Sodium | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  24-hour Urine Sodium will assessed using ISE indirect for 24 hour urine collection with (mmol/24Hr) units of measures.The reference range is 40-220 mmol/24hr. Higher than 220 mmol/24hr is not recommended.
Change 24-hour Urine Potassium | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  24-hour Urine Potassium will assessed using ISE indirect for 24 hour urine collection with (mmol/24Hr) units of measures. The reference range 25-125 mmol/24hr. Higher than 125 mmol/24hr is not recommended.
Change Diastolic Blood Pressure | Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (Five week post-intervention)
  Diastolic Blood Pressure will be assessed using CARESCAPE DINAMAP technology digital blood pressure monitor model V100, BP assessor will obtain three BP measures in the right arm after the participant has been sitting quietly for 5 min. An average of the 3 measures is recorded.The recommended Diastolic Blood Pressure lower of 80 mm Hg.

CONTACTS AND LOCATIONS:
Overall Officials: Boon How Chew, PhD, Study Chair — Universiti Putra Malaysia
Locations (1):
- Al Sawad, Ayat, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Ayat Ali AS, Lim SK, Tang LY, Rashid AA, Chew BH. The effectiveness of nurse-led self-management support program for people with chronic kidney disease stage 3-4 (CKD-NLSM): Study protocol for a randomized controlled trial. Sci Prog. 2021 Apr-Jun;104(2):368504211026159. doi: 10.1177/00368504211026159. PMID 34143698